CLINICAL TRIAL: NCT06121115
Title: Norepinephrine Administration Through a Midline Catheter in an Intermediate Care Unit - a Retrospective Study of Complications and Patient Outcomes
Brief Title: Norepinephrine Administration Through a Midline Catheter in an Intermediate Care Unit
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-06476
Record Dates: First submitted 2023-10-03; First posted 2023-11-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Septic Shock; Norepinephrine Adverse Reaction; Hypotension and Shock
Keywords: vasopressor; norepinephrine; septic shock; midline catheter; thrombosis; extravasation; catheter-related bloodstream infection
MeSH Terms: conditions — Shock, Septic; Hypotension; Shock; Thrombosis | interventions — Norepinephrine; Vasoconstrictor Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine administered in midline catheter according to clinical routine
  Other Names: Vasopressors

SUMMARY:
This is a single-center study retrospectively evaluating a local clinical routine to administer norepinephrine in midline catheters, with regard to complications and patient outcomes

DETAILED DESCRIPTION:
Se attached study protocol

ELIGIBILITY:
Inclusion Criteria:

* Administration of norepinephrine in a midline catheter in an intermediary care unit
* In Skåne university hospital
* From 2019 to 2023-03-31

Exclusion Criteria:

* Patients who have actively disabled review of their electronic medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are critically ill patients in need of vasopressors, primarily with septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a major complication of norepinephrine administration in midline | day 30
  extravasation of norepinephrine, midline-associated bloodstream infection, thrombosis

SECONDARY OUTCOMES:
Proportion of patients with a minor complication of norepinephrine administration in midline | day 30
  infiltration, occlusion of midline, dislodgement, leakage, other
Proportion of patients receiving a CVC after midline | day 30
  Has the patient received central line after midline placement
Proportion of patients with different intermediary care unit outcomes | day 30
  Where did the patient go after intermediary care? discharged / escalated to the ICU / deceased

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Torisson, PhD, Principal Investigator — Region Skåne
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karlsson H, Afrasiabi A, Ohlsson M, Mansson V, Hartman H, Torisson G. Treating shock with norepinephrine administered in midline catheters in an intermediary care unit: a retrospective cohort study. BMJ Open. 2024 Dec 30;14(12):e091311. doi: 10.1136/bmjopen-2024-091311. PMID 39806688

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT06121115/Prot_SAP_000.pdf